CLINICAL TRIAL: NCT02474186
Title: Phase II Study of Chemo-Radiation-Induced Abscopal Effect in Metastatic Breast Cancer and in Other Metastatic Sites of Solid Tumors
Brief Title: Phase II Study for Solid Metastatic Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-58
Record Dates: First submitted 2015-06-03; First posted 2015-06-17 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; Solid Tumor
Keywords: breast; cancer; metastatic; breast cancer; metastatic breast cancer; radiation; radiotherapy; radiation therapy; abscopal; abscopal effect; T-cell; GM-CSF; anti-tumor; immune; immune response; capecitabine; xeloda; taxol; paclitaxel; other solid metastatic tumor
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Radiotherapy; Capecitabine; Paclitaxel; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiation therapy (Experimental): Patients with metastatic breast cancer and other metastatic solid tumors receiving single-agent chemotherapy will receive 3.5 Gy/fraction to a total dose of 35 Gy/10 fractions over 2 weeks with concurrent systemic therapy
  Systemic agents are either capecitabine (Xeloda), paclitaxel, docitaxel or taxol
  Interventions: Radiation: Radiation therapy; Drug: Xeloda; Drug: paclitaxel

INTERVENTIONS:
Radiation: Radiation therapy — Patients with metastatic breast cancer and other metastatic solid tumors receiving single-agent chemotherapy will receive 3.5 Gy/fraction to a total dose of 35 Gy/10 fractions over 2 weeks with concurrent systemic therapy
  Other Names: Radiotherapy
Drug: Xeloda — chemotherapy agent daily for two weeks
  Other Names: capecitabine
Drug: paclitaxel — chemotherapy agent weekly for two weeks
  Other Names: docetaxel; taxol

SUMMARY:
1. To induce immunity-mediated tumor response outside the radiation field (abscopal effect) after chemo-radiation of a metastatic site in metastatic breast cancer patients.
2. To monitor the induction of a T cell response.
3. To explore the role of PET scanning to assess tumor responses/abscopal effect.

DETAILED DESCRIPTION:
1. To induce immunity-mediated tumor response outside the radiation field (abscopal effect) after chemo-radiation of a metastatic site in a pilot study of metastatic breast and other metastatic solid tumors.
2. To monitor the induction of a T cell response in patients with metastatic breast cancer.
3. To explore the role of PET scanning to assess tumor response/abscopal effect.

Eligible are women with metastatic breast cancer and patients with other metastatic solid tumors who have achieved stable disease or have disease progression after systemic therapy and have at least three separate measurable sites of disease. Extent of metastatic disease is recorded both at CT and PET scanning. Radiation is given during systemic therapy to one of the lesions, 35 Gy in ten fractions over a two week interval, conformally to maximally spare normal tissue. GM-CSF treatment is given daily for fourteen days. At day 22 radiation is re-started and the same radiation dose is delivered to a second metastatic site, again with GM-CSF. Abscopal response is evaluated by assessing clinical and PET response in the non-irradiated measurable metastatic sites. A Phase II clinical trial based on an optimum two-stage Phase II Simon design is used to conduct this pilot study. Ten patients will be treated in Stage one; if there are no abscopal responses, the trial will be terminated. If there are one or more abscopal responses in Stage One, the trial will proceed to enroll an additional 19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed breast cancer or other cancer which is persistent and metastatic or recurrent and metastatic.
* Patients with a history of treatment for other prior malignancy will be eligible, provided they remain disease-free > 2 years after initial treatment, or were treated for non-melanoma skin cancer, or in situ cervical cancer.
* Patients must have at least 3 distinct measurable metastatic sites at least 1 cm of larger in their largest diameter.
* Age >18 years.
* ECOG performance status <2 (Karnofsky >50%).
* Life expectancy > 3 months.

Exclusion Criteria:

* Patients who have had immunotherapy within 4 weeks prior to entering the study.
* Patients who have had prior allergic reaction to GM-CSF
* Patients on steroid therapy or other immunosuppressive therapy.
* Patients undergoing therapy with other investigational agents.
* Patients with known brain metastases can be included in this clinical trial but brain lesions are not eligible as target or non target lesion.
* Uncontrolled inter-current illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, myocardial infarction within the past 6 months, unstable angina pectoris, or unstable cardiac arrhythmia requiring assessment for clinical intervention.

Ages: 19 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2003-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with an abscopal response assessed at 7-8 weeks after the initiation of treatment. | week 7- week 8

SECONDARY OUTCOMES:
The number of participants with adverse events from the date of enrollment until 12 years from the opening of the study. | year 0 - year 12
The proportion of patients alive with abscopal responses from the date of enrollment until date of death from any cause, assessed up to 12 years from the opening of the study. | year 0- year 12

CONTACTS AND LOCATIONS:
Overall Officials: Encouse Golden, M.D., Ph.D., Principal Investigator — NYU School of Medicine

REFERENCES:
- [Derived] Golden EB, Chhabra A, Chachoua A, Adams S, Donach M, Fenton-Kerimian M, Friedman K, Ponzo F, Babb JS, Goldberg J, Demaria S, Formenti SC. Local radiotherapy and granulocyte-macrophage colony-stimulating factor to generate abscopal responses in patients with metastatic solid tumours: a proof-of-principle trial. Lancet Oncol. 2015 Jul;16(7):795-803. doi: 10.1016/S1470-2045(15)00054-6. Epub 2015 Jun 18. PMID 26095785